CLINICAL TRIAL: NCT05451173
Title: Combining an Immune Checkpoint Inhibitor With SBRT or Hypo-fractionated RT in the Treatment of Stage I-III NSCLC: an Exploratory Study on Radiation Dose and Treatment Efficacy.
Brief Title: Combining ICI With SBRT or HypoFrx-RT for ES NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexander Chi (Other)
Responsible Party: Sponsor-Investigator, Alexander Chi, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF 2022-2-1042
Record Dates: First submitted 2022-06-29; First posted 2022-07-11 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer; Non-small Cell Carcinoma; Non-small Cell Lung Cancer Stage I; Non-small Cell Lung Cancer Stage II; Non-small Cell Lung Cancer Stage III
Keywords: NSCLC, Stereotactic body radiotherapy, SBRT, Hypofractionated, Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Radiation Dose Hypofractionation; durvalumab

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): SBRT to be delivered with concurrent and adjuvant anti-PD-(L)1 immune checkpoint inhibitor.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Durvalumab
- Cohort B (Experimental): Hypo-fractionated radiotherapy to be delivered with concurrent and adjuvant anti-PD-(L)1 immune checkpoint inhibitor.
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — An ablative dose of radiation is delivered to the primary tumor target over 1-2 week.
  Other Names: SBRT
  Arms: Cohort A
Radiation: Hypofractionated radiotherapy — Hypofractionated radiotherapy is delivered to the primary tumor and any involved lymph node target(s) over 3 weeks.
  Other Names: HypoFrx-RT
  Arms: Cohort B
Drug: Durvalumab — an anti-PD-(L)1 immune checkpoint inhibitor is administered concurrently and adjuvantly with radiotherapy.

SUMMARY:
This study will explore the best dose of radiation to be used when treating stage I-III non-small cell lung cancer (NSCLC) with stereotactic body radiation therapy (SBRT) or hypo-fractionated radiotherapy (HypoFrx-RT) that is delivered in combination with an immune checkpoint inhibitor. Treatments with SBRT or HypoFrx-RT for locally confined NSCLC show positive response which may be further augmented when they are combined with an immune checkpoint inhibitor. Currently, it is not understood what radiation dose is most suitable for such combined treatments and their clinical efficacy in the treatment of early stage (ES) NSCLC. Therefore, this study can help researchers gain insight into what a safe and effective SBRT or HypoFrx-RT dose will be when such radiotherapeutic approaches are combined with concurrent and adjuvant administration of an immune checkpoint inhibitor in the treatment of ES NSCLC.

DETAILED DESCRIPTION:
Patients will be assigned to Cohort A or Cohort B based on tumor stage (AJCC 8th Ed.).

Cohort A: cT1-T3, N0, M0 (selected cT1, No, M0)

Cohort B: cT4, N0, M0; cT1-4, N1-3, M0

Phase I:

This portion of the study will utilize a standard 3 + 3 phase I design with three patients enrolled per radiation dose level in each cohort. Enrollment in the two cohorts is independent from one another. In both cohorts, an anti-PD-(L)1 immune checkpoint inhibitor will be given concurrently and adjuvantly with radiotherapy for approximately 1 year.

The radiation dose escalation for each cohort is listed below:

Cohort A (SBRT):

(Optional): 8 Gy x 5 daily fractions

Level 1: 9 Gy x 5 daily fractions

Level 2: 10 Gy x 5 daily fractions

Level 3: 11 Gy x 5 daily fractions

Cohort B (HypoFrx-RT):

(Optional): 3 Gy x 15 daily fractions

Level 1: 3.5 Gy x 15 daily fractions

Level 2: 4 Gy x 15 daily fractions

DLTs will be based on events occurring during the course of radiotherapy.

Concurrent administration of an immune checkpoint inhibitor is defined as:

An anti-PD-(L)1 immune checkpoint inhibitor administered with standard dosing (Durvalumab: 1500 mg every 4 weeks) given within 5 days prior to the beginning of radiotherapy.

Adjuvant administration of an immune checkpoint inhibitor is defined as:

An anti-PD-(L)1 immune checkpoint inhibitor administered with standard dosing (Durvalumab: 1500 mg every 4 weeks) for approximately 1 year or until progression or other discontinuation criteria are met.

Phase II:

Once a maximum tolerated dose (MTD) is defined in each cohort, this dose will be used as the only radiation dose in each corresponding cohort in the phase II portion of this study. Dosing regimen of the immune checkpoint inhibitor will remain the same as that used in the phase I portion of this study.

For this protocol, patients will be followed up to 2 years after the last dose of immune checkpoint inhibitor is administered.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria

1. Informed Consent
2. Stage I-III NSCLC per AJCC 8th. ed.
3. Tumor PD-L1 expression ≥1% preferred
4. Tumor sample submission
5. Tumor staging prior to registration
6. Age ≥ 18 years
7. WHO/ECOG PS of 0, 1, or 2
8. Life expectancy ≥12 weeks
9. Adequate organ or bone marrow function
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.

Exclusion Criteria:

Key Exclusion Criteria

1. Mixed small cell and non-small cell lung cancer histology
2. Definitive clinical or radiologic evidence of metastatic disease
3. Patients who received systemic therapy for the current cancer prior to enrollment
4. Thoracic radiotherapy within 5 years with exceptions
5. Major surgery within 28 days prior to enrollment with exception
6. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody
7. History of another primary malignancy with exceptions
8. History of idiopathic pulmonary fibrosis, any pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on chest PET/CT or CT scan
9. Active or prior documented autoimmune disease with exceptions
10. History of primary immunodeficiency
11. History of allogenic organ or tissue transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 2 years
  MTD in cohort A and cohort B, respectively.
The incidence of any adverse events that is >= grade 3 | 2 years
  Adverse events will be graded according to CTCAE v.5.0
Progression-free survival (PFS) | 2 years
  PFS is defined as free from any disease progression or death after combined treatment for NSCLC.

SECONDARY OUTCOMES:
Local control | 2 years
  To report the local control rate along with the rate of regional control and distant metastasis after combined treatment for NSCLC.
Overall survival (OS) | 2 years
  To report OS after combined treatment
Quality of Life (QoL) | 2 years
  To determine the QoL pertaining to any cancer patients before and after treatment using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire, Core 30 (EORTC QLQ-C30) scales.
Quality of Life (QoL), Lung cancer specific | 2 years
  To determine the QoL before and after treatment using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire that is specific to lung cancer patients, the Lung Cancer 29(LC 29) scoring scales.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chi, MD, Study Chair — Capital Medical University
Locations (1):
- Capital Medical University Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No